CLINICAL TRIAL: NCT04288063
Title: Chemical Fingerprints of Skeletal Muscle Health in Children With Type 1 Diabetes
Brief Title: Skeletal Muscle Health in Children With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00104288
Record Dates: First submitted 2020-02-26; First posted 2020-02-27 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early onset T1D children: 25 young, prepubertal and very early pubertal (Tanner stages 1 and 2) children (13 females and 12 males) with early onset T1D

SUMMARY:
The purpose of this research study is to find out if Type 1 Diabetes (T1D) affects skeletal muscle health and if we can improve glycemic control by improving skeletal muscle health. Participants in this study will have a blood sample and a urine sample collected after taking a single dose of a nontoxic chemical called D3-creatine. Their body composition will be measured by a scale like device. Parents of participating children will also be asked to complete a food and activity questionnaire.

Participants will be in the study for roughly 12 to 24 months. Enrollment will begin once participant signs the consent form. At the 12 month follow-up visit participants will be asked to wear a Garmin physical activity monitor and use the Garmin Connect mobile app for a period of up to 12 months and take a one time Muscle Strength Measurement test.

The greatest risks of this study include the possibility of loss of confidentiality.

DETAILED DESCRIPTION:
Physical Activity Monitor:

This research will look at the relationship of physical activity on skeletal muscle health, by using a Physical Activity Monitor (Garmin vívofit 3): At the 12 month follow-up visit study participant will be asked to wear a Garmin physical activity monitor and use the Garmin Connect mobile app for a period of up to 12 months. The Garmin Connect app will be downloaded onto the parent or guardian's smartphone or tablet. The study team will create a unique study-specific Duke email (e.g. SMHparticipantXXX@duke.edu) and an assign a unique password for each participant. Passwords will be assigned in accordance with applicable Duke Health password security policy requirements. This email address and password will be used solely for account creation and will not be used for communication. No personal information will be used in the study-specific email or password. Study participants are advised to limit personal identifiers entered into mobile applications/third party software only to those that you wish to voluntarily share with others. Study participant is under no obligation to participate in this phase of the study, as is the case with all research, this sub-study is 100% voluntary.

Measurement of Muscle Strength:

Upper and lower body strength will be measured using tools that give the researchers a snapshot of the strength in specific muscle groups. Participant will be asked to grip or pinch or push or pull against a device that measures the force they generate when doing these tasks, to measure their strength. In addition to muscle strength testing we will be measuring functional endurance by having participant walk for 6 minutes to see how far they can walk in 6 minutes. These measurements will be taken by a physical therapist in coordination with regularly scheduled appointments.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 3 months (defined by American Diabetes Association criteria, with glutamic acid decarboxylase, islet cell or insulin autoantibodies, and insulin requirement.
* Age ≥6 to 11 (inclusive) years of age
* Tanner stage 1 and 2 (pre-pubertal and early pubertal) to minimize pubertal effects
* Normal weight, overweight and obese children with weight maintenance (no recent significant weight loss or gain). Normal weight will be defined as a BMI between the 5th and 85th percentile; overweight will be defined as a BMI at or above the 85th percentile and below the 95th percentile, obesity will be defined as a BMI at or above the 95th percentile for children of the same age and sex
* Mobile Phone needed for Activity Monitoring device App

Exclusion Criteria:

* Current or recent (within the past month) use of medications affecting IR (oral or inhaled steroids, metformin, thiazolidinediones, or atypical antipsychotics)
* Genetic syndrome causing diabetes
* Untreated hypothyroidism
* Proteinuria, which could affect the metabolomic profiling.
* Anemia or hemoglobinopathies that could affect HbA1c levels,
* Underweight or recent weight loss.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cohort will consist of 25 young, prepubertal and very early pubertal (Tanner stages 1 and 2) children (13 females and 12 males) with early onset T1D
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-11-19 (Actual)

PRIMARY OUTCOMES:
Change in muscle mass as measured by D3 creatinine dilution method | Baseline, 1 year

SECONDARY OUTCOMES:
Physical Activity | Up to 1 year
  Continuously monitor physical activity of step count using a mobile device (Garmin).
Endurance | Baseline (Sub-study)
  Measured by a 6 minute walk test of physical activity endurance
Muscle Strength | Baseline (Sub-study)
  Determined by use of dynamometry measurements

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Gumus Balikcioglu, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No